CLINICAL TRIAL: NCT06998199
Title: Effects Of Dual Task Balance Exercises Versus Vestibular Stimulation On Balance Control and Gross Motor Coordination In Children With Down Syndrome
Brief Title: Dual Task Balance Exercises and Vestibular Stimulation for Children With Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/24/0748
Record Dates: First submitted 2025-04-24; First posted 2025-05-31 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Down Syndrome
Keywords: Down syndrome; balance control; Vestibular stimulation; Dual Task balance exercise; gross motor coordination
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Intervention Model Description: A Randomized clinical trial performed, in which 26 Down Syndrome children with the age of 7 to 14 years will be taken randomly after screening and meeting inclusion criteria.
  Children will be divided in two groups. Group 1 will receive Dual task balance exercises and Group 2 will receive Vestibular stimulations. Both groups will receive total of 16 sessions, 2 sessions per week for 8 weeks. Each session lasted 30-45 min on average. Pre values were taken at 1st week and post values will be taken after 8th week of intervention to measure the effects of both therapies.
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols and possible efforts will be put to mask the both group about the treatment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual Task Balance exercise group (Experimental): Experimental: Dual Task Balance exercise group Clinical experimental: For group -A dual task balance exercise at least lasted 30-45 min on average . 15 minutes for dual task exercise and 30 min for routine physical therapy.Patients will receive total of 16 sessions, 2 sessions per week for 8 weeks.
  Interventions: Other: Dual Task Balance Exercise
- Vestibular Stimulation group (Active Comparator): Active Comparator: VS Group Clinical experimental: For group B VS lasted at least 30-45 min on average . 15 minutes for VS and 30 min for routine physical therapy.Patients will receive total of 16 sessions, 2 sessions per week for 8 weeks.
  Interventions: Other: Vestibular Stimulation

INTERVENTIONS:
Other: Dual Task Balance Exercise — The content of the DT training is summarized below with 30 minutes of routine PT. Participants will receive total of 16 sessions, 2 sessions per week for 8 weeks.
  1. Walking 3 m on hard/soft ground while performing a motor task (carrying an empty box) and then combined with a cognitive task (saying the names of some fruits and vegetables),
  2. Sitting on a Pilates ball for 1 min with eyes open/closed while performing a motor task (arms flexed to 90 degrees) and then combined with a cognitive task (saying the names of friends)
  3)2-feet Jumping forward with both feet for 3 m while performing a motor task (carrying an empty box) then with a cognitive task (naming the colors in the room)
  4)Standing on one leg for 30 s while arms abducted to 90 degrees and then combined with a cognitive task (saying the names of relatives)
  5)Sit-to-stand using a stool 15 repetitions with a motor task (carrying an empty box) and then with a cognitive task (saying the names vegetables etc)
  Arms: Dual Task Balance exercise group
Other: Vestibular Stimulation — The child will place in sitting position on the swing and his hands grasping the ropes at the sides then the therapist stand behind him and begin pushing the platform in fast and jerky movement in back and front, side to side and in spinning directions with the child trying to maintain his balance in all different directions. The subject will receive pushing for each direction for five minutes; the total mechanical vestibular session duration was 15 minutes with 30 minutes of routine physical therapy. Participants will receive total of 16 sessions, 2 sessions per week for 8 weeks.
  Arms: Vestibular Stimulation group

SUMMARY:
Children with Down syndrome experience balance and postural control issues due to neuromuscular defects and face several impairments. For the improvement we will take 26 children with Down syndrome, age between 7 to 14 years will be randomly assign into two groups.

Group A will perform Dual Task Balance exercises and group B will perform Vestibular Stimulation exercises along routine physical therapy.All the data will be collected from Rabia Welfare Hospital Lahore by using Pediatric Balance Scale, Time Up and Go test and KTK test.The duration of study will be 10 months. Data will be analyzed through SPSS version 25.00.

DETAILED DESCRIPTION:
Down syndrome is a genetic disorder experience balance issues due to neuromuscular defects which present with several impairments such as hypotonic, ligament laxity, decreased muscle strength, insufficient muscular co-contraction, inadequate postural control, intellectual disabilities, sensory integration difficulties and disturbed proprioception. The current study will be randomized clinical trial, data will be collected from Rabia Welfare Hospital Lahore. The study will include 26 patients equally divided into two groups and randomly allocated. Inclusion criteria for the study will include patients diagnosed with Down syndrome, age between 7 to 14 years(both genders), able to understand instructions and command necessary for intervention and children which able to stand momently but with history of frequent falling during walking. Patients with Atlanto axial instability, Cardiopulmonary, Orthopedic and Neurological problems, cognitive impairment that interferes with communication, BMI of ≥30 kg/m2 and children which actively participating in sports will be excluded.Group A will perform Dual Task Balance exercises and group B will perform Vestibular Stimulation exercises along routine physical therapy.Both groups will receive total of 16 sessions, 2 sessions per week for 8 weeks. Each session lasted 30-45 min on average.Then evaluate both groups on follow up.Before and after intervention period, balance and gross motor coordination will be assessed by Pediatric Balance Scale, Time Up and Go test and KTK test. The reliability and validity of tools mentioned. Data collection will be done before and after the intervention. Data will be analyzed through SPSS version 25.00.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Down syndrome.
* Age between 7 to 14 years.
* Both the genders were included.
* Able to talk and comprehend instructions & command.
* Children which able to stand momently but with history of frequent falling during walking

Exclusion Criteria:

* Child with Atlanto axial instability.
* Uncontrolled cardiopulmonary problems.
* Body mass index (BMI) of ≥30 kg/m2.
* Children with orthopedic problems and affecting gait.
* Cognitive impairment that interferes with communication.
* Neurological problems.
* Children which actively participating in sports

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2025-04-18 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2025-06-16 (Actual)

PRIMARY OUTCOMES:
The Pediatric Balance Scale | Baseline, 1st week and 8th week
  The Pediatric Balance Scale (PBS), a modified version of Berg's Balance Scale, was designed to assess balance in school-aged children with mild to severe motor deficits. The scale consists of 14 items that are scored from 0 points (lowest function) to 4 points (highest function) with a maximum score of 56 points. Reliability testing performed with a sample of 20 children ages 5-15 years old with mild to moderate motor impairments showed good test-retest reliability (ICC=0.998) and good inter rater reliability (ICC=0.997)
Timed up and go test | Baseline, 1st week and 8th week
  The 'timed up and go' test (TUG) is a simple, quick and widely used clinical performance based measure of lower extremity function, mobility and fall risk.
  1. Begin by having the patient sit back in a standard arm chair and identify a line 3 meters, or 10 feet away, on the floor.
  2. On the word "Go," begin timing.
  3. Stop timing after patient sits back down.
  4. Record the time. The TUG has demonstrated good test-retest reliability (ICC 0.80-0.99), validity, and sensitivity to change. It has a moderate correlation with fall risk
Körperkoordinationstest für Kinder (KTK) | Baseline, 1st week and 8th week
  The Körperkoordinationstest für Kinder (KTK), also known as the Body Coordination Test for Children to measure gross motor coordination in children aged 5 to 15 years. The KTK consists of four subtests: walking backward on balance beams of varying widths, jumping sideways with both feet together, moving sideways on boxes, and hopping for height on one leg which takes 15 minutes per child. The results from the four tasks are used to calculate a Motor Quotient (MQ). A score below an MQ of 85 is typically considered indicative of motor difficulties. KTK showed acceptable construct validity, indeed, the test-retest for the raw score on the test protocol detected a reliability coefficient of 0.97, and for each item, reliability coefficients ranged from (0.80 to 0.96).

CONTACTS AND LOCATIONS:
Overall Officials: Amina Shafaqut, MS-PPT, Principal Investigator — Riphah International University
Locations (1):
- Rabia Welfare Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buyukcelik NM, Yigit S, Turhan B. An investigation of the effects of dual-task balance exercises on balance, functional status and dual-task performance in children with Down syndrome. Dev Neurorehabil. 2023 Jul;26(5):320-327. doi: 10.1080/17518423.2023.2233031. Epub 2023 Jul 4. PMID 37403442